CLINICAL TRIAL: NCT04533646
Title: Comparison of Meal-Time Dosing of Rapid Acting Insulin Using Carbohydrate Counting vs. Fixed Doses Utilizing Continuous Glucose Monitoring In Patients With Cystic Fibrosis Related Diabetes
Brief Title: Comparison of Meal-Time Dosing of Insulin in Cystic Fibrosis Related Diabetes
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Jagdeesh Ullal (Other)
Collaborators: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor-Investigator, Jagdeesh Ullal, Clinical Associate Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY20060197
Record Dates: First submitted 2020-08-23; First posted 2020-08-31 (Actual); Results first posted 2025-03-19 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Cystic Fibrosis-related Diabetes
MeSH Terms: interventions — Insulin

STUDY DESIGN:
Intervention Model Description: This study design involves a within-subjects comparison using a sequential cross over that occurs over a 2-week time frame. During the first seven days of wear, the participants will be asked to dose their mealtime rapid-acting insulin by fixed-dose, and the next seven days, participants will be asked to dose their mealtime rapid-acting insulin by carbohydrate counting. After the 14 days, participants will return their continuous glucose monitor (CGM) devices for analysis and interpretation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Fixed Dosing, Followed by Carbohydrate Counting (Experimental): Dosing of premeal insulin with fixed doses
  Interventions: Drug: Insulin; Device: Continuous glucose monitor (CGM)

INTERVENTIONS:
Drug: Insulin — Participants will be asked to dose insulin during the first week using fixed doses. During the second week of the study, participants will dose insulin based on carbohydrate counting. Blood sugar control will be compared between the 2 weeks to determine the outcomes of the study.
Device: Continuous glucose monitor (CGM) — Participants will be required to wear a CGM to measure glucose trends

SUMMARY:
The aim of this study is to assess the utility of CGMs to determine the optimal method to dose meal-time insulin. The investigators will examine glucose excursions in patients with CF who will dose meal-time rapid-acting insulin by carbohydrate counting versus fixed-dose rapid-acting insulin. The carbohydrate ratio and fixed doses will be determined by existing doses, total daily insulin doses, body weight, and insulin sensitivity along with predisposition to hypoglycemia. Bolus insulin dosing is an important part of CFRD management due to the high nutritional demands of these patients. If dosed incorrectly, this could lead to marked hyperglycemia and could worsen nutritional status due to urinary glucose losses. In this project, the investigators will perform a within-subjects' comparison of the 2 standard methods of meal-time rapid-acting insulin dosing.

DETAILED DESCRIPTION:
Background and Introduction Cystic fibrosis-related diabetes (CFRD) is the most common extra-pulmonary comorbidity in patients with cystic fibrosis (CF). CFRD is also associated with an accelerated decline in pulmonary function, increased pulmonary exacerbations, and increased mortality. Continuous glucose monitoring (CGM) involves the use of a small disposable sensor sited in the subcutaneous interstitial fluid that makes frequent glucose measurements. There is data suggesting that the Medtronic iPro continuous glucose monitors (CGM) can predict hemoglobin a1c levels in patients with CFRD.

The aim of this study is to assess the utility of CGMs to determine the optimal method to dose meal-time insulin. The investigators will examine glucose excursions in patients with CF who will dose meal-time rapid-acting insulin by carbohydrate counting versus fixed-dose rapid-acting insulin. The carbohydrate ratio and fixed doses will be determined by existing doses, total daily insulin doses, body weight, and insulin sensitivity along with predisposition to hypoglycemia. Bolus insulin dosing is an important part of CFRD management due to the high nutritional demands of these patients. If dosed incorrectly, this could lead to marked hyperglycemia and could worsen nutritional status due to urinary glucose losses. In this project, the investigators will perform a within-subjects' comparison of the 2 standard methods of meal-time rapid-acting insulin dosing.

Hypothesis:

1. Postprandial interstitial fluid glucose levels in participants who utilize carbohydrate counting to dose mealtime rapid-acting insulin will have improved control as defined as the area under the curve and time in target compared to participants who used fixed-dose mealtime insulin
2. Participants who utilize carbohydrate counting will have fewer hypoglycemia events compared to participants who use fixed-dose meal-time insulin

Specific Aims:

1. To compare within-subject glucose excursions defined as the percentage of time in target glucose level, percentage of glucose in target, and peak postprandial glucose with fixed insulin dosing versus carbohydrate count based insulin dosing.
2. To compare the frequency and duration of hypoglycemia (defined as the daily, weekly, and average duration of the event) between insulin delivery methods described above.
3. To test the use of 'rule of 500' for carb counting estimation in patients with CFRD
4. To compare the effect of two methods of rapid-acting insulin delivery on fasting glycemia

ELIGIBILITY:
Inclusion Criteria:

* Age >18 age of years
* Diagnosis of cystic fibrosis related diabetes
* Using basal bolus insulin
* Cystic Fibrosis with Lung Transplantation

Exclusion Criteria:

* Use of continuous glucose monitors
* Patient unable to check fingerstick blood sugars

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2020-09-15 (Actual); Primary Completion 2023-07-31 (Actual); Study Completion 2025-09-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jagdeesh Ullal, MD, Principal Investigator — University of Pittsburgh Medical Center
Locations (1):
- University of Pittsburgh Medical Center, Center for Diabetes and Endocrinology, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study subjects were recruited from the Cystic Fibrosis Diabetes Clinic. The study was started on 9-15-2020 and concluded on 07-31-2023.
Pre-assignment Details: Study subjects served as their own controls. There was no wash out or run-in period.
Period: Fixed Insulin Dosing (7 Days)
Arm/Group | Fixed Dosing, Followed by Carbohydrate Counting
Started | 13
Completed | 8
Not Completed | 5
Period: Carbohydrate Counting ( 7 Days)
Arm/Group | Fixed Dosing, Followed by Carbohydrate Counting
Started | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Fixed Dosing, Followed by Carbohydrate Counting
Number analyzed (Participants) | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 12
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 8
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 12
  More than one race | 1
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 13
Baseline weight [Mean (Standard Deviation); unit: pounds] | 152 (9)

OUTCOME MEASURES:

1. Primary Outcome: Time in Target
Description: Measurement of percentage of time in target of glucose level
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: percentage of time in range
Arm/Group | Fixed Dosing, Followed by Carbohydrate Counting
Number analyzed (Participants) | 8
percentage of time in range
  Fixed Dose | 67 (5.9)
  Carb Counting | 68 (0.4)
Statistical Analysis 1: Comparison: Fixed Dosing, Followed by Carbohydrate Counting; Test type: Other; p < 0.01, Means testing; Mean Difference (Net) = 1.1; comparison of means test was performed

2. Secondary Outcome: Hypoglycemia
Description: To determine the time spent in hypoglycemia as defined as blood sugar under 70 mg/dl
Time Frame: 2 weeks
Measure: Mean (Standard Deviation); unit: minutes
Groups:
- Fixed Dosing Followed by Carbohydrate Counting: Dosing of premeal insulin with fixed dose insulin followed by carbohydrate counting
  Insulin: Participants will be asked to dose insulin during the first week using fixed doses. During the second week of the study, participants will dose insulin based on carbohydrate counting. Blood sugar control will be compared between the two weeks to determine the study's outcomes.
  Continuous glucose monitor (CGM): Participants will be required to wear a CGM to measure glucose trends
Arm/Group | Fixed Dosing Followed by Carbohydrate Counting
Number analyzed (Participants) | 8
minutes
  Fixed dose | 134 (54)
  Carb Counting | 112 (57)

ADVERSE EVENTS:
Time Frame: 2 weeks
Groups:
- Fixed Dosing: Dosing of premeal insulin with fixed doses
  Insulin: Participants will be asked to dose insulin during the first week using fixed doses.
  Continuous glucose monitor (CGM): Participants will be required to wear a CGM to measure glucose trends
- Carb Counting: Dosing of premeal insulin with carb counting
  Insulin: During the second week of the study, participants will dose insulin based on carbohydrate counting.
  Continuous glucose monitor (CGM): Participants will be required to wear a CGM to measure glucose trends
Arm/Group | Fixed Dosing | Carb Counting
All-Cause Mortality (participants affected / at risk) | 0/13 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/13 | 0/8
Other Adverse Events (participants affected / at risk) | 0/13 | 0/8

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-08-03): https://cdn.clinicaltrials.gov/large-docs/46/NCT04533646/Prot_SAP_000.pdf